CLINICAL TRIAL: NCT04847349
Title: Live Microbials to Boost Anti-SARS-CoV-2 Immunity Clinical Trial (Live BASIC Trial)
Brief Title: Live Microbials to Boost Anti-Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Immunity Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Vault Health, Inc. (Unknown); Danisco USA Inc. (Unknown)
Responsible Party: Principal Investigator, Daniel B. Horton, MD, MSCE, Assistant Professor of Pediatrics and Epidemiology, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Pro2021000186
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Covid19
Keywords: Probiotics
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Live microbial (Probiotic) consortium OL-1, standard dose (Experimental): Combination of a standard dose of live microbials (probiotics) taken as a capsule once per day with breakfast for 21 days. Capsules should not be consumed with hot drinks or alcohol.
  Interventions: Dietary Supplement: OL-1, standard dose
- Live microbial (Probiotic) consortium OL-1, high dose (Experimental): Combination of a high dose of live microbials (probiotics) taken as a capsule once per day with breakfast for 21 days. Capsules should not be consumed with hot drinks or alcohol.
  Interventions: Dietary Supplement: OL-1, high dose
- Placebo for live microbial (probiotic) consortium (Placebo Comparator): Capsule containing inactive ingredients such as a product of potato starch (maltodextrin), but no probiotics, taken once per day with breakfast for 21 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: OL-1, standard dose — The live microbial components have been present in the food supply, have a long history of safe use in foods, and are already marketed in the United States.
  Arms: Live microbial (Probiotic) consortium OL-1, standard dose
Dietary Supplement: OL-1, high dose — The live microbial components have been present in the food supply, have a long history of safe use in foods, and are already marketed in the United States.
  Arms: Live microbial (Probiotic) consortium OL-1, high dose
Dietary Supplement: Placebo — Capsule containing inactive ingredients such as a product of potato starch (maltodextrin), but no probiotics.
  Arms: Placebo for live microbial (probiotic) consortium

SUMMARY:
This pilot double-blind randomized controlled trial will test the preliminary efficacy of two doses of a combination of live microbials (probiotics) given to boost the immunity of unvaccinated persons previously infected with SARS-CoV-2.

DETAILED DESCRIPTION:
This pilot double-blind randomized controlled trial will test the preliminary efficacy of two doses (a standard dose and a high dose) of a combination of live microbials (probiotics), currently marketed in food (including products labeled as dietary supplements), given daily for 21 days to boost the immunity of unvaccinated, generally healthy persons ages 18-60 with prior confirmed SARS-CoV-2 infection. Data collected will include demographics, comorbidities, medications, information about prior SARS-CoV-2 infection, and self-reported symptoms and adverse events (AEs). Biospecimens (saliva, nasal wash, blood, and stool) will be collected at baseline and days 21 and 42 for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (any gender, ages 18 to 60 years old) in good general health, based on medical history
* SARS-CoV-2 infection >4 months prior confirmed by a positive polymerase chain reaction (PCR) or antigen test
* Body mass index (BMI) of 18.5-39.9 kg/m2
* Agreement to comply with the protocol and study restrictions
* Access to internet in addition to willingness and ability to use web-based questionnaires
* Available for all study visits
* English-speaking

Exclusion Criteria:

* Recent infection with coronavirus disease-2019 (COVID-19) (newly positive PCR or antigen test within prior 4 months)
* Prior receipt of antibody therapies (convalescent or monoclonal) towards COVID-19
* Prior receipt of vaccines against COVID-19
* Prior or current participation in a clinical trial of vaccines against COVID-19
* Scheduled to receive a vaccine against COVID-19 in the following month
* Regular use of any live microbial (probiotic) supplements
* Any acute or chronic respiratory tract disease besides mild to moderate asthma
* Any diagnosed immunodeficiency
* Current use of immunosuppressive drugs
* Any diagnosis of chronic gut disease, such as inflammatory bowel disease or irritable bowel syndrome
* Pregnancy or breastfeeding
* Recent use of antibiotics
* Current addiction to alcohol, drugs, or medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change in titer of serum anti-SARS-CoV-2 immunoglobulin G (IgG) | between baseline and day 21 (day 1 is the first day of taking the investigational product)

SECONDARY OUTCOMES:
Change in the titer of serum anti-SARS-CoV-2 IgG | between baseline and day 42
Change in the titer of serum anti-SARS-CoV-2 neutralizing antibody | between baseline and days 21 and 42
Change in the titer of serum and nasal anti-SARS-CoV-2 immunoglobulin A (IgA) antibody | between baseline and days 21 and 42
In-vitro changes in cytokine release in response to stimulation of peripheral blood mononuclear cells with SARS-CoV-2 peptides | between baseline and days 21 and 42
Serum cytokine levels | between baseline and days 21 and 42
Adverse events | up to 10 weeks
Change in any baseline symptoms from prior SARS-CoV-2 infection | up to 6 weeks
New (repeat) SARS-CoV-2 infections | up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Horton, MD, MSCE, Principal Investigator — Rutgers University
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Saliva, nasal rinse, blood samples, and stool samples collected will be used for the purposes of this research.
  After information that could identify consenting participants has been removed, de-identified information and left over biospecimens collected for this research may be used by or distributed to the study funder (Danisco USA Inc.) or to investigators for other research without obtaining additional informed consent. Personal identifying details, such as name and date of birth, will not be shared without participants' additional permission.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared after enrollment and data analysis are completed.

REFERENCES:
- [Derived] Horton DB, Ukey R, Madhvi A, Andrews T, Parmar V, Reilly N, Makela SM, Peterson J, Hustad L, Wong G, Barrett ES, Bruiners N, Carson JL, Getz K, Greenberg P, Iizuka A, Roy J, Pastuszak AW, Lehtinen MJ, Blaser MJ, Panettieri RA Jr, Gennaro ML. Live microbials to boost Anti-SARS-CoV-2 immunity clinical trial (Live BASIC trial): a triple-blind randomized controlled trial. Infection. 2025 Nov 26. doi: 10.1007/s15010-025-02697-4. Online ahead of print. PMID 41299123